CLINICAL TRIAL: NCT02814786
Title: In Vivo Dynamic Evaluation of Ankle Joint and Muscle Mechanics in Children With Spastic Equinus Deformity Due to Cerebral Palsy: Implications for Recurrent Equinus.
Brief Title: Dynamic Evaluation of Ankle Joint and Muscle Mechanics in Children With Spastic Equinus Deformity Due to Cerebral Palsy
Acronym: EQUINUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of inclusion
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RB15-159 EQUINUS
Record Dates: First submitted 2016-02-10; First posted 2016-06-28 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Equinus Deformity
MeSH Terms: conditions — Equinus Deformity | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Equinus cohort (Experimental): 15 childrens who have a fixed equinus defined as a fixed limitation of dorsiflexion inferior to 0°.
  Interventions: MRI scanner and gait analysis
  Interventions: Radiation: MRI scanner; Other: Gait analysis
- Control cohort (Experimental): In this cohort, there will be 15 childrens with age and gender matched to equinus cohort and with no history of lower limb musculo-skeletal injury in past 6 months.
  Interventions: MRI scanner and gait analysis
  Interventions: Radiation: MRI scanner; Other: Gait analysis

INTERVENTIONS:
Radiation: MRI scanner — This examination is divided in 2 parts:
  * Passive movement: after placing the ankle joint in the fixture, each child will be asked to relax the lower limb musculature and then the fixture will be cyclically moved by a technician at a speed which does not trigger spasticity.
  * Active movement: no technician will be present and children will be asked to perform voluntary plantar-dorsiflexion between the extreme positions on the beat of the metronome.
  Other Names: MRI data on pediatric ankle joint
Other: Gait analysis — For gait evaluation, each child will undergo a lower limb gait analysis in a motion analysis laboratory equipped with Camera system and 4 AMTI force plates Sixteen reflective markers will be placed on the lower limbs. Each child will walk bare foot and gait will be recorded during each of five 10-meter trials. A velocity of 1 m/s (+/- 10%) will be imposed using a stop watch in order to eliminate the influence of velocity on gait kinematics and kinematics while comparing across subjects. Each child will be allowed to walk for 5 minutes after attaching the reflective markers and before recording the gait data. In addition to the joint kinematics, joint powers and moments will be computed using an inverse dynamics method.
  Other Names: Gait evaluation

SUMMARY:
This research will lead to the first evaluation of intrinsic and dynamic joint and muscle mechanics of equinus in cerebral palsy. It would provide a direct cause and effect relationship between equinus and bone deformity. Mechanical insights to the pathophysiology of the targeted muscles will lead to better understanding and, thus, to a better medical and surgical management of equinus deformity. Secondary aim will provide an important insight whether key gait parameters can be exclusively relied upon for surgical treatment planning and evaluation. In a medium-term perspective, depending upon the results of this study, dynamic MRI of the ankle joint may serve as a guiding tool for fixed equinus surgery in case of cerebral palsy.

DETAILED DESCRIPTION:
Equinus is the most common deformity in children with cerebral palsy. Spastic equinus is typically defined as the inability to dorsa-flex the foot above plantigrade, with the hindfoot in neutral position and the knee in extended position. Approximately 90% of the deformities in cerebral palsy occur in the ankle and foot region alone with the incidence of equinus being around 75%. Spastic equinus exhibits poor muscle control and muscle weakness around ankle and foot, resulting in bone deformities and gait abnormalities. Non-operative conservative management of equinus is typically undertaken up until 8 years in order to prevent recurrent equinus or overcorrection by avoiding high-growth phase of child's development for surgical intervention. Despite these precautions, long term follow-up studies report up to 48% of recurrence rate post-surgery. Recurrence surgery not only increases the economic burden on the society but also has a debilitating impact on children and their families. Previous research is focused on extrinsic risk factors such as CP type, demographic parameters, and clinical gait parameters for surgical recurrence and none assessed the dynamic impact of intrinsic bone deformity on ankle joint and muscle mechanics. A primary reason for this recurrence could be a lack of understanding of bone deformity that might be forcing the child to adapt altered ankle joint and muscle mechanics (bone kinematics, cartilage contact parameters, muscle strain) during dynamic activities. In fact, the surgical treatment of fixed equinus does not consider any bone corrections and focus on muscle release or lengthening only. Being a dynamic pathology, it is critical to understand the in vivo effect of weak ankle joint musculature on joint mechanics and the resultant bone deformity. However, no such efforts have been made so far in the literature. With the advent of technology, researchers have developed and validated dynamic magnetic resonance imaging techniques to analyze in vivo muscle and joint mechanics. Processing this data enables researchers to analytically track bones without having to identify specific points or anatomical landmarks and thus provides the ability to track muscle motion as well as skeletal motion. Thus properties such as bone kinematics, cartilage contact mechanics, musculotendon moment arms, muscle strain and tendon strain are available from these analyses. These techniques can be successfully employed in equinus research to evaluate ankle joint and muscle mechanics in vivo.

ELIGIBILITY:
Equinus cohort inclusion criteria:

* children between 7 and 14 years old
* with unilateral CP and GMFCS score of I or II
* with the presence of fixed equinus defined as a fixed limitation of dorsiflexion inferior to 0°

Control cohort inclusion criteria:

* age and gender matched to equinus cohort
* no history of lower limb musculo-skeletal injury in past 6 months
* no history of lower limb musculoskeletal surgery in past six months
* no contraindications to MRI

Equinus cohort exclusion criteria:

* history of lower limb musculo-skeletal surgery
* botulinum toxin injection in past 6 months
* contraindications to MRI
* Uncooperative patient who refused to sign the informed consent
* Patient unable to understand the protocol, under guardianship
* Patients not affiliated to the Social Security.

Control cohort exclusion criteria:

* Uncooperative patient who refused to sign the informed consent
* Patient unable to understand the protocol, under guardianship
* Patients not affiliated to the Social Security.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Talocrural joint flexion, pronation, and internal rotations | One year
  Talocrural (talus relative to tibia) joint rotations and translations will be compared between two cohorts.
Subtalar joint flexion, pronation, and internal rotations | one year
  Subtalar (calcaneus relative to talus) joint rotations and translations will be compared between two cohorts.
Achilles tendon moment arm (MAAT) | one year
  MAAT is defined as a perpendicular 3D distance between Achilles' tendon line of action and the Medial-lateral Calcaneal axis. Using calcaneal kinematics, MAAT value for each time frame will be quantified and compared between two cohorts.

SECONDARY OUTCOMES:
Ankle joint kinematics (joint angles) during walking | one year
  Walking gait parameters (ankle, knee, and hip joint angles) will be correlated with primary outcome measures
Knee joint kinematics (joint angles) during walking | one year
  Walking gait parameters (ankle, knee, and hip joint angles) will be correlated with primary outcome measures
Hip joint kinematics (joint angles) during walking | one year
  Walking gait parameters (ankle, knee, and hip joint angles) will be correlated with primary outcome measures
Talocrural joint contact area | one year
  Joint contact mechanics measures and will be compared between cohorts.
Talocrural joint contact centroid location | one year
  Joint contact mechanics measures and will be compared between cohorts.
Subtalar joint contact area | one year
  Joint contact mechanics measures and will be compared between cohorts.
Subtalar joint contact centroid location | one year
  Joint contact mechanics measures and will be compared between cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makki K, Borotikar B, Garetier M, Acosta O, Brochard S, Ben Salem D, Rousseau F. 4D in vivo quantification of ankle joint space width using dynamic MRI. Annu Int Conf IEEE Eng Med Biol Soc. 2019 Jul;2019:2115-2118. doi: 10.1109/EMBC.2019.8856687. PMID 31946318
- [Background] Cheng, Y., Bailly, R., Borotikar, B., Scavinner-Dorval, C., Fouquet, B., Salem, D. B., ... & Rousseau, F. (2023, April). Morphological analysis of ankle shorts bones of children with cerebral palsy: a comparative study. In Medical Imaging 2023: Image Processing (Vol. 12464, pp. 584-588). SPIE.
- [Background] Scavinner-Dorval, C., Bailly, R., Borotikar, B., Brochard, S., Salem, D. B., & Rousseau, F. (2024, April). Analysis of disentangled representation learning for high-resolution dynamic MRI synthesis. In Medical Imaging 2024: Image Processing (Vol. 12926, pp. 694-699). SPIE